CLINICAL TRIAL: NCT03964597
Title: Objective Measurements of Lens Opacification After Intravitreal Injections (MOC-IVT)
Brief Title: Objective Measurements of Lens Opacification After Intravitreal Injections
Acronym: MOC-IVT
Status: Withdrawn | Type: Observational
Why Stopped: Study abandoned before any submission (foreseeable organizational difficulties)
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: EBA_2019_9
Record Dates: First submitted 2019-05-24; First posted 2019-05-28 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Lens Opacification; Intravitreal Injections (IVT)
Keywords: Cataract; objective scatter index (OSI); average lens density (ALD)
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Measurement of lens opacification — Measurement of OSI and ALD at inclusion and during post-IVT follow-up visits to M3, M6, and M12, +/- M18, +/- M24 and +/- M30.

SUMMARY:
The main hypothesis is the opacification of the lens would be increase by the IVT.

The opacification of the lens can be objectived by :

* the objective scatter index (OSI) on the OQAS device
* the average lens density (ALD) on the IOLMaster device.

Eligible patients will be followed at least 12 months after in intravitreal injection and the opacification of their lens is regularly controlled with OSI and ALD.

The objective is to study the dynamics of lens opacification in IVT-treated eyes evaluated by OSI for at least 1 year.

ELIGIBILITY:
Inclusion criteria:

* An indication of an intravenous injection of a dexamethasone 700 μg (Ozurdex®) or anti-VEGF for at least one of the two eyes for macular edema or neovessels linked to DMLA, retinal venous occlusion, diabetic macular edema or posterior uveitis
* Phake patient, at least of the injected eye

Exclusion criteria:

- Pseudophakia of the injected eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an indication for intravitreal injection (IVT) for medical condition.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Value of the OSI (Objective Scatter Index) in one year of follow-up after IVT | 12 months

IPD SHARING:
Plan to Share IPD: No